CLINICAL TRIAL: NCT06734702
Title: Neoadjuvant Immunotherapy Plus Chemotherapy Followed by Concurrent Chemoradiotherapy and Consolidative Immunotherapy Compared With Concurrent Chemoradiotherapy and Consolidative Immunotherapy in Locally Advanced Non-small Cell Lung Cancer: A Randomized, Phase III Controlled Study
Brief Title: Neoadjuvant Immunotherapy Plus Chemotherapy Followed by Concurrent Chemoradiotherapy and Consolidative Immunotherapy for Locally Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10124
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Neoadjuvant Therapy; Concurrent Chemoradiotherapy; Immunotherapy; Locally Advanced Non-Small Cell Lung Cancer
Keywords: Neoadjuvant therapy; Concurrent Chemoradiotherapy; Immunotherapy; Locally Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group A (Experimental): Patients will receive neoadjuvant chemo-immunotherapy, hypo-RT and concurrent chemotherapy, followed by consolidative immunotherapy for a maximum duration of 12 months.
  Interventions: Drug: Neoadjuvant therapy; Radiation: Hypo-RT and concurrent chemotherapy; Drug: Consolidative immunotherapy
- Study group B (Experimental): Patients will receive neoadjuvant chemo-immunotherapy, CFRT and concurrent chemotherapy, followed by consolidative immunotherapy for a maximum duration of 12 months.
  Interventions: Drug: Neoadjuvant therapy; Radiation: CFRT and concurrent chemotherapy; Drug: Consolidative immunotherapy
- Control group (Active Comparator): CFRT and concurrent chemotherapy, followed by consolidative immunotherapy for a maximum duration of 12 months.
  Interventions: Radiation: CFRT and concurrent chemotherapy; Drug: Consolidative immunotherapy

INTERVENTIONS:
Drug: Neoadjuvant therapy — The neoadjuvant regimen prior to radiotherapy consists of albumin-bound paclitaxel 260 mg/m², cisplatin 75 mg/m², and tislelizumab 200 mg, administered every 3 weeks.
  Arms: Study group A; Study group B
Radiation: Hypo-RT and concurrent chemotherapy — Definitive dose of hypofractionated thoracic radiotherapy with concurrent chemotherapy
  Arms: Study group A
Radiation: CFRT and concurrent chemotherapy — Definitive dose of conventionally fractionated thoracic radiotherapy with concurrent chemotherapy
  Arms: Control group; Study group B
Drug: Consolidative immunotherapy — Following the completion of chemoradiotherapy, Tislelizumab consolidation therapy will be administered based on treatment efficacy and the patient's physical condition, for a total duration of 1 year, starting 1-2 months after chemoradiotherapy.

SUMMARY:
Consolidative immunotherapy following concurrent chemoradiotherapy, based on the PACIFIC trial, has become the standard treatment for locally advanced non-small cell lung cancer (LANSCLC), leading to a 5-year survival rate of over 40%. The optimal timing of radiotherapy combined with immunotherapy still requires further exploration. This phase III, randomized controlled clinical trial is to investigate the efficacy and safety of neoadjuvant immuno-chemotherapy followed by concurrent chemoradiotherapy and consolidative immunotherapy, compared with concurrent chemoradiotherapy and consolidative immunotherapy in LANSCLC patients.

DETAILED DESCRIPTION:
This phase III, randomized controlled trial aims to investigate the efficacy and safety of neoadjuvant immuno-chemotherapy followed by concurrent chemoradiotherapy and consolidative immunotherapy, compared with concurrent chemoradiotherapy and consolidative immunotherapy in LANSCLC patients. Patients will be randomized in a 2:2:1 ratio to the following three groups: Group A: Patients will receive neoadjuvant chemo-immunotherapy. After neoadjuvant therapy, they will undergo hypofractionated radiotherapy (hypo-RT) and concurrent chemotherapy, followed by consolidative immunotherapy for a maximum duration of 12 months. (2) Group B: Patients will receive neoadjuvant chemo-immunotherapy. After neoadjuvant therapy, they will undergo conventionally fractionated radiotherapy (CFRT) and concurrent chemotherapy, followed by consolidative immunotherapy for a maximum duration of 12 months. (3) Group C: Patients will receive CFRT and concurrent chemotherapy, followed by consolidative immunotherapy for a maximum duration of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed and Dated Informed Consent: Written informed consent must be provided prior to any study procedures, with the consent form signed and dated by the participant.
* Age Range: Male or female patients aged 18 to 75 years.
* Diagnosis: Patients must have locally advanced, unresectable (stage III) non-small cell lung cancer (NSCLC), with histological or cytological confirmation of the diagnosis.
* Previous Treatment: Patients must not have received prior chemotherapy, radiotherapy, surgery, targeted therapy, or immunotherapy.
* Tumor Sample Requirement: Tumor tissue samples must be provided, and they should be sufficient for analysis. The samples must be unstained and archived.
* Life Expectancy: Patients must have an expected survival of at least 12 weeks.
* Performance Status (PS): The patient's WHO Performance Status (PS) must be 0 or 1.
* Pregnancy Testing: Postmenopausal women, or women who have had a negative urine or serum pregnancy test within 14 days before the study medication (HCG sensitivity ≥ 25 IU/L or equivalent).
* Breastfeeding: Women must not be breastfeeding.
* Women of childbearing potential (WOCBP) must agree to use contraception during the study treatment period and for 5 months after the last dose of the investigational drug (i.e., 30 days [ovulation cycle] + approximately 5 half-lives of the study drug).
* Men who have sexual relations with WOCBP must agree to use contraception during the study treatment period and for 7 months after the last dose of the investigational drug (i.e., 90 days [sperm renewal cycle] + approximately 5 half-lives of the study drug).
* Males with no sperm production are exempt from contraception requirements. WOCBP who are not sexually active are exempt from contraception but must still undergo pregnancy testing as outlined above.
* Organ and Bone Marrow Function: The following laboratory parameters must be met:

Forced expiratory volume in 1 second (FEV1) ≥ 800 mL Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L Platelets ≥ 100 × 10⁹/L Hemoglobin ≥ 9.0 g/dL Calculated creatinine clearance using the Cockcroft-Gault formula ≥ 50 mL/min Serum bilirubin ≤ 1.5 × upper limit of normal (ULN) AST and ALT ≤ 2.5 × ULN

Exclusion Criteria:

* Patients meeting any of the following criteria should not be enrolled in the study:
* Concurrent participation in another clinical trial, except for observational (non-interventional) studies.
* Histological subtype of mixed small-cell and non-small-cell lung cancer. Use of immunosuppressive drugs within 28 days before treatment, except for intranasal or inhaled corticosteroids at physiological doses or systemic corticosteroids ≤10 mg/day of prednisone or equivalent.
* Prior treatment with anti-PD-1 or anti-PD-L1 antibodies.
* Major surgery within 4 weeks prior to enrollment (excluding procedures for vascular access).
* History or active autoimmune diseases within the past two years.
* Active or a history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of organ transplantation requiring immunosuppressive therapy.
* Average corrected QT interval (QTc) ≥470 ms calculated from three ECG cycles using the Bazett formula.
* Uncontrolled comorbidities, including but not limited to: Persistent or active infections. Symptomatic congestive heart failure. Poorly controlled hypertension. Unstable angina. Cardiac arrhythmias. Active peptic ulcer disease or gastritis. Active bleeding disorders. Hepatitis C or HIV infection. HBsAg-positive patients with HBV DNA >500 IU/mL. Mental or social conditions that may limit adherence to study requirements or compromise the ability to provide informed consent.
* Known history of tuberculosis.
* Receipt of a live attenuated vaccine within 30 days before study initiation or planned during the study period.
* History of another primary malignancy within the past 5 years, except for adequately treated basal or squamous cell carcinoma of the skin or in situ cervical cancer.
* Pregnancy, breastfeeding, or not using effective contraception (for men and women of reproductive potential).

Patients in the experimental group should not proceed to concurrent chemoradiotherapy if any of the following criteria are met:

* Presence of distant metastases.
* Locoregional progression making definitive concurrent chemoradiotherapy unfeasible due to normal tissue dose constraints (assessed by the radiation oncologist).
* WHO performance status score of 2-4.
* Impaired organ or bone marrow function, including:

Forced expiratory volume in 1 second (FEV1) <800 mL. Absolute neutrophil count (ANC) <1.5 × 10⁹/L. Platelets <100 × 10⁹/L. Hemoglobin <9.0 g/dL. Creatinine clearance (Cockcroft-Gault formula) <50 mL/min. Serum bilirubin >1.5 × upper limit of normal (ULN). AST and ALT >2.5 × ULN.

- Patient withdrawal from the study.

Patients should not proceed to consolidation immunotherapy if any of the following criteria are met:

* Disease progression during concurrent chemoradiotherapy.
* Use of immunosuppressive drugs within 28 days before the first dose of tislelizumab, except for physiological doses of intranasal or inhaled corticosteroids or systemic corticosteroids ≤10 mg/day of prednisone or equivalent. Use of corticosteroids to manage chemoradiotherapy-related toxicity is permitted.
* Persistent unresolved CTCAE grade >2 toxicities from prior chemoradiotherapy.
* Grade ≥2 pneumonitis resulting from prior chemoradiotherapy.
* Any prior grade ≥3 immune-related adverse event (irAE) or unresolved irAE > grade 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2028-11-29 (Estimated); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival rate | 18-months
  PFS measures the time from the start of treatment until the disease progresses or the patient dies from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1-2 months after treatment
  ORR refers to the proportion of patients who experience complete response (CR) and partial response (PR)
Overall survival (OS) | 2 years
  OS is the time from the start of treatment until death from any cause.
Failure patterns | 2 years
  Failure patterns describe the pattern of disease progression or treatment failure, such as local recurrence or distant metastases
Safety: Adverse Events of Grade 2 or Higher | 1 years after treatment
  Safety endpoints assess the frequency and severity of treatment-related adverse events (side effects). Adverse events are graded on a scale from 1 to 5, with grade 2 and above indicating more significant side effects that may require medical intervention or treatment modifications.
Quality of life assessed by Quality of Life Core 30 | 1 years after treatment
  Patient-reported quality of life measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Higher scores on functioning scales indicate better functioning, while higher scores on symptom scales indicate more severe symptoms.
Quality of life assessed by Quality of Life LC13 | 1 years after treatment
  Patient-reported quality of life measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-LC13). Higher scores on functioning scales indicate better functioning, while higher scores on symptom scales indicate more severe symptoms.
The percentage of patients who are eligible for consolidative immunotherapy following chemoradiotherapy | 1 year
  The percentage of patients who are eligible for consolidative immunotherapy following chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Deenen MJ, Dewit L, Boot H, Beijnen JH, Schellens JH, Cats A. Simultaneous integrated boost-intensity modulated radiation therapy with concomitant capecitabine and mitomycin C for locally advanced anal carcinoma: a phase 1 study. Int J Radiat Oncol Biol Phys. 2013 Apr 1;85(5):e201-7. doi: 10.1016/j.ijrobp.2012.12.008. PMID 23517808
- [Background] Wu B, McNutt T, Zahurak M, Simari P, Pang D, Taylor R, Sanguineti G. Fully automated simultaneous integrated boosted-intensity modulated radiation therapy treatment planning is feasible for head-and-neck cancer: a prospective clinical study. Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):e647-53. doi: 10.1016/j.ijrobp.2012.06.047. Epub 2012 Aug 3. PMID 22867890
- [Background] Franceschini D, Paiar F, Meattini I, Agresti B, Pasquetti EM, Greto D, Bonomo P, Marrazzo L, Casati M, Livi L, Biti G. Simultaneous integrated boost-intensity-modulated radiotherapy in head and neck cancer. Laryngoscope. 2013 Dec;123(12):E97-103. doi: 10.1002/lary.24257. Epub 2013 Jun 26. PMID 23775348
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Liao ZX, Komaki RR, Thames HD Jr, Liu HH, Tucker SL, Mohan R, Martel MK, Wei X, Yang K, Kim ES, Blumenschein G, Hong WK, Cox JD. Influence of technologic advances on outcomes in patients with unresectable, locally advanced non-small-cell lung cancer receiving concomitant chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):775-81. doi: 10.1016/j.ijrobp.2009.02.032. Epub 2009 Jun 8. PMID 19515503
- [Background] Provencio M, Nadal E, Insa A, Garcia-Campelo MR, Casal-Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Casarrubios M, Salas Anton C, Parra ER, Wistuba I, Calvo V, Laza-Briviesca R, Romero A, Massuti B, Cruz-Bermudez A. Neoadjuvant chemotherapy and nivolumab in resectable non-small-cell lung cancer (NADIM): an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Nov;21(11):1413-1422. doi: 10.1016/S1470-2045(20)30453-8. Epub 2020 Sep 24. PMID 32979984
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Durm GA, Jabbour SK, Althouse SK, Liu Z, Sadiq AA, Zon RT, Jalal SI, Kloecker GH, Williamson MJ, Reckamp KL, Langdon RM, Kio EA, Gentzler RD, Adesunloye BA, Harb WA, Walling RV, Titzer ML, Hanna NH. A phase 2 trial of consolidation pembrolizumab following concurrent chemoradiation for patients with unresectable stage III non-small cell lung cancer: Hoosier Cancer Research Network LUN 14-179. Cancer. 2020 Oct 1;126(19):4353-4361. doi: 10.1002/cncr.33083. Epub 2020 Jul 22. PMID 32697352
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Sacco PC, Maione P, Guida C, Gridelli C. The Combination of New Immunotherapy and Radiotherapy: A N ew Potential Treatment for Locally Advanced Non-Small Cell Lung Cancer. Curr Clin Pharmacol. 2017;12(1):4-10. doi: 10.2174/1574884711666161201123439. PMID 27908252
- [Background] Wang Y, Deng W, Li N, Neri S, Sharma A, Jiang W, Lin SH. Combining Immunotherapy and Radiotherapy for Cancer Treatment: Current Challenges and Future Directions. Front Pharmacol. 2018 Mar 5;9:185. doi: 10.3389/fphar.2018.00185. eCollection 2018. PMID 29556198